CLINICAL TRIAL: NCT03579836
Title: A Single Center, Open-label, Non-comparative, Phase I/II Clinical Trial to Assess the MTD, Safety and Efficacy of BEY1107 in Monotherapy and in Combination with Gemcitabine in Patient with Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Evaluation of Safety and Efficacy in BEY1107 in Monotherapy Gemcitabine Combination in Patient with Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeyondBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BEY-2018-01
Record Dates: First submitted 2018-06-08; First posted 2018-07-09 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced or Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase I-1 (#4 Cohort) (Experimental): BEY1107 monotherapy, 4 Cohorts, 4 weeks (administered on a 3-week-on and 1-week-off)
  Interventions: Drug: BEY1107
- Phase I-2 (#3 Cohort) (Experimental): BEY1107 in combination with Gemcitabine, 3 Cohorts, 4 weeks (administered on a 3-week-on and 1-week-off)
  Interventions: Drug: BEY1107; Combination Product: Gemcitabine
- Phase II (#1 Cohort) (Experimental): BEY1107 in combination with Gemcitabine, 6 Cycles / 24 weeks (administered on a 3-week-on and 1-week-off)
  Interventions: Drug: BEY1107; Combination Product: Gemcitabine

INTERVENTIONS:
Drug: BEY1107 — Take orally with water once a day on a 3-weeks-on (21 days) continuously and 1-week-off (7 days) schedule.
Combination Product: Gemcitabine — Administer 1,000 mg/m2 of Gemcitabine intravenously for 30 minutes on Day 1, 8, 15 and 1-week-off (7days) schedule.
  Arms: Phase I-2 (#3 Cohort); Phase II (#1 Cohort)

SUMMARY:
This study is a single center, open-label, non-comparative, phase I/II clinical trial to assess the maximum tolerated dose (MTD), safety and efficacy of BEY1107 in monotherapy and in combination with gemcitabine in patient With locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
The key purpose of the main part of the study is to assess the MTD, safety and efficacy of BEY1107 as monotherapy and combination therapy for locally advanced and/or metastatic pancreatic cancer. The main purpose of the safety lead-in (dose-finding) part of the study is to determine the safety and tolerability of BEY1107, to determine the MTD.

Patient will receive BEY1107 for 4 weeks in monotherapy for each cohort (administered in a 3-weeks-on / 1-week-off) during Phase I-1 trial.

At next stage, patient will receive BEY1107 with gemcitabine for 4weeks in phase I-2 trial.

Final stage, patient will receive BEY1107 with gemcitabine for 24weeks in phase II trial.

Blood samples will be collected for safety, pharmacokinetic and biomarker analysis. Archival of fresh biopsy tissue will also be collected for biomarker analysis.

ELIGIBILITY:
Inclusion criteria :

1. Histologically or Cytologically confirmed with pancreatic ductal adenocarcinoma or undifferentiated carcinoma of the pancreas
2. At lease one measurable lesion according to RECIST v.1.1
3. Eastern Cooperative Oncology Group (ECOG) 0,1 or 2
4. Over 12 weeks of Life expectancy
5. Adequate Bone marrow, Renal and Liver function at screening

Exclusion criteria :

1. A patient who has treatment history with locally advanced and/or metastatic pancreatic cancer
2. Major surgery history at screening
3. Uncontrolled brain metastasis evidence
4. Active bacterial infection patients
5. Malignant tumor other than basal cell carcinoma, cervix carcinoma in situ and papillary thyroid cancer
6. expected Pregnant or breast-feeding patients
7. HIV, Active hepatitis B or C infection
8. A patient who has hypersensitivity with BEY1107 or Gemcitabine

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-05-14 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MTD & Safety assessment (Phase I) | 0
DCR(Disease Control Rate) in combination therapy of BEY1107 and Gemcitabine (Phase II) | 0

SECONDARY OUTCOMES:
AUC in BEY1107 monotherapy and Gemcitabine combination (Phase I) | 0
Cmax in BEY1107 monotherapy and Gemcitabine combination (Phase I) | 0
DCR(Disease Control Rate) in BEY1107 monotherapy and Gemcitabine combination (Phase I) | 0
ORR(Objective Response Rate) in BEY1107 and Gemcitabine combination (Phase II) | 0
Number of subjects with Adverse events in BEY1107 and Gemcitabine combination (Phase II) | 0

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No